CLINICAL TRIAL: NCT04246372
Title: Safety and Efficacy of Tofacitinib for Immune Skin Conditions in Down Syndrome
Brief Title: Tofacitinib for Immune Skin Conditions in Down Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1362; R33AR077495 (NIH)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome; Alopecia Areata; Atopic Dermatitis / Eczema; Hidradenitis Suppurativa; Vitiligo; Psoriasis
Keywords: Interferon; Autoimmunity; Down syndrome; Skin disorder; JAK inhibitor; Inflammation; JAK/STAT; Dermatology
MeSH Terms: conditions — Down Syndrome; Alopecia Areata; Dermatitis, Atopic; Eczema; Hidradenitis Suppurativa; Vitiligo; Psoriasis; Autoimmune Diseases; Skin Diseases; Inflammation | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: All participants will receive the investigational product, Tofacitinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- On Treatment (Experimental): Tofacitinib 5mg oral tablets twice daily for 16 weeks
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Treatment with oral Tofacitinib for immune mediated skin conditions in adults with Down syndrome
  Other Names: Xeljanz

SUMMARY:
People with Down syndrome (DS) display widespread immune dysregulation, including several immune skin conditions. This study hypothesizes that pharmacological inhibition of the increased interferon (IFN) signaling seen in DS is safe and could improve associated skin conditions.

The study evaluates the safety and efficacy treatment with Tofacitinib, an FDA-approved drug known to block IFN signaling, in adolescents and adults with DS and an autoimmune and/or autoinflammatory skin condition. Investigators will also measure the impact of interferon inhibition on a variety of molecular markers, as well as the cognitive abilities and quality of life of participants.

DETAILED DESCRIPTION:
Trisomy 21 (T21) is the most common human chromosomal disorder, occurring in ~1/700 live births, leading to the condition known as Down syndrome (DS). Importantly, people with DS display widespread immune dysregulation and over half of adults with T21 are affected by one or more autoimmune conditions, including several immune skin conditions. The driving hypothesis for this study is that hyperactivation of interferon (IFN) signaling leads to myriad immune-driven diseases and immunological phenotypes in people with DS, and that pharmacological inhibition of IFN signaling could have multidimensional therapeutic benefits in this population.

This study utilizes Tofacitinib, an FDA-approved drug known to block IFN signaling and several accompanying inflammatory pathways, to reduce IFN signaling in DS and to measure its effects via multidimensional endpoints. Previous studies and current clinical trials indicate that Janus kinase (JAK) inhibitors, such as Tofacitinib, can block inflammatory pathways and may have beneficial effects on immune skin conditions. Further, inhibition of chronically active IFN signaling in DS with Tofacitinib may attenuate other core drivers of immune dysregulation, leading to improvements in other immune diseases and conditions common to DS that are potentially driven by inflammation, such as cognitive deficits. Investigators will test these hypotheses using a battery of immune and molecular assessments, as well as cognitive testing and quality of life measures. This clinical trial evaluates adolescent and adult participants with DS during eight study visits over an approximate five month period.

Specific Aims:

1. To define the safety profile of JAK inhibition in people with DS,
2. To determine the impact of JAK inhibition on the immune dysregulation caused by trisomy 21,
3. To define the impact of JAK inhibition on immune skin conditions in DS, and
4. To characterize the impact of JAK inhibition on cognition and quality of life in DS.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with DS between 12 and 50 years of age who weigh at least 40 kg.
* Diagnosis of at least one active immune skin condition, including but not limited to:

  1. Moderate-to-severe atopic dermatitis
  2. Alopecia areata affecting at least 25% of the scalp
  3. Moderate-to-severe hidradenitis suppurativa
  4. Moderate-to-severe psoriasis
  5. Moderate-to-severe vitiligo.
* Be willing to avoid pregnancy or fathering children.
* Must present with a study partner or legal guardian who can complete, or assist with completing, study materials as appropriate.

Exclusion Criteria

* Weigh less than 40 kg.
* Pregnancy or breast feeding.
* No study partner or legal guardian.
* Vaccination with live attenuated virus within six weeks of inclusion in the study or planned during the study.
* Clinically significant chronic or active viral infection including but not limited to HIV, hepatitis, CMV, EBV, HSV.
* Severe renal impairment.
* History of malignant solid tumor cancer within five years prior to study entry or where there is current evidence of recurrent or metastatic disease.
* Poor venous access not allowing repeated blood tests or non-compliance with venipuncture requirements.
* Prior treatment with a JAK inhibitor or with an investigational agent, device, or procedure within 21 days of enrollment.
* Concomitant treatment with other immunosuppressants (e.g. corticosteroids, methotrexate) or strong CP3A4 or CYP2C19 inhibitors or inducers (e.g. ketoconazole, fluconazole).
* Known allergies, hypersensitivity, or intolerance to Tofacitinib.
* History of thrombotic disorder.
* Superficial skin infection within 2 weeks of inclusion in the study.
* History of disseminated herpes zoster, disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
* Intravenous antimicrobial therapy within 3 months of inclusion in the study.
* Oral antimicrobials within 2 weeks of inclusion in the study.
* Participants may be excluded for other unforeseen reasons at the study doctor's discretion.
* Unable to provide assent in cases where informed consent is obtained from other authorized representative.
* Kidney transplant within the last two years
* Any history of heart attack or stroke.
* Any history of lymphoma.
* Past or current smokers.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Espinosa, PhD, Principal Investigator — Linda Crnic Institute, University of Colorado Anschutz Medical Campus
Locations (1):
- Linda Crnic Institute for Down Syndrome, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available for all primary outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available upon publication in a peer-reviewed journal.
Access Criteria: Data access requests will be reviewed by the sponsor-investigator and collaborators.

REFERENCES:
- [Background] Rachubinski AL, Estrada BE, Norris D, Dunnick CA, Boldrick JC, Espinosa JM. Janus kinase inhibition in Down syndrome: 2 cases of therapeutic benefit for alopecia areata. JAAD Case Rep. 2019 Apr 5;5(4):365-367. doi: 10.1016/j.jdcr.2019.02.007. eCollection 2019 Apr. No abstract available. PMID 31008170
- [Background] Pham AT, Rachubinski AL, Enriquez-Estrada B, Worek K, Griffith M, Espinosa JM. JAK inhibition for treatment of psoriatic arthritis in Down syndrome. Rheumatology (Oxford). 2021 Sep 1;60(9):e309-e311. doi: 10.1093/rheumatology/keab203. No abstract available. PMID 33630031
- [Derived] Rachubinski AL, Wallace E, Gurnee E, Enriquez-Estrada BA, Worek KR, Smith KP, Araya P, Waugh KA, Granrath RE, Britton E, Lyford HR, Donovan MG, Eduthan NP, Hill AA, Martin B, Sullivan KD, Patel L, Fidler DJ, Galbraith MD, Dunnick CA, Norris DA, Espinosa JM. JAK inhibition decreases the autoimmune burden in Down syndrome. Elife. 2024 Dec 31;13:RP99323. doi: 10.7554/eLife.99323. PMID 39737640
- [Derived] Rachubinski AL, Wallace E, Gurnee E, Estrada BAE, Worek KR, Smith KP, Araya P, Waugh KA, Granrath RE, Britton E, Lyford HR, Donovan MG, Eduthan NP, Hill AA, Martin B, Sullivan KD, Patel L, Fidler DJ, Galbraith MD, Dunnick CA, Norris DA, Espinosa JM. JAK inhibition decreases the autoimmune burden in Down syndrome. medRxiv [Preprint]. 2024 Oct 16:2024.06.13.24308783. doi: 10.1101/2024.06.13.24308783. PMID 38946973
- See also: The Crnic Institute Human Trisome Project — http://www.trisome.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On Treatment
Started | 47
Completed | 42
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Total number of participants who completed Baseline visit and were considered to be enrolled (n=47).
  All enrolled participants are represented in Safety Outcome Measure.
  As the Primary Outcome Measure for Whole Blood Transcriptome Interferon (IFN) Score is based on the change between Baseline and 16 weeks, a Baseline Measure for this Outcome is based on the 39 completed participants analyzed for this Primary Outcome based on medication compliance and sample availability.
Arm/Group | On Treatment
Number analyzed (Participants) | 47
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 22 [18.2 to 25.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 5
  Unknown or Not Reported | 0
Whole Blood Transcriptome Interferon (IFN) Score [Median (Inter-Quartile Range); unit: IFN score] — The Interferon Score is a composite molecular measure used to quantify activation of the interferon signaling pathway. Interferon Scores are calculated by summing standardized expression (i.e. (expression value - mean) / standard deviation) of a predefined panel of 16 interferon-stimulated genes, measured by RNA-sequencing of whole blood samples. The resulting composite value provides an integrated measure of interferon pathway activity, with higher scores indicating greater pathway activation. No clinical relevance threshold has been established. Population: Median IFN score with IQR was calculated for 39 participants who completed 16 weeks.
  IFN score
    number analyzed (Participants) | 39
    (all) | 5.28 [1.71 to 8.85]

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events (SAE) Definitely Related to Tofacitinib Treatment.
Description: Safety as measured by the number of serious adverse events definitely related to tofacitinib treatment.
Time Frame: Baseline to 16 weeks
Population: All participants who attended Baseline appointment.
Measure: Number; unit: Serious Adverse Events
Arm/Group | On Treatment
Number analyzed (Participants) | 47
Serious Adverse Events | 0

2. Primary Outcome: Change in Whole Blood Transcriptome Interferon (IFN) Score
Description: The Interferon Score is a composite molecular measure used to quantify activation of the interferon signaling pathway. Interferon Scores are calculated by summing standardized expression (i.e. (expression value - mean) / standard deviation) of a predefined panel of 16 interferon-stimulated genes, measured by RNA-sequencing of whole blood samples. The resulting composite value provides an integrated measure of interferon pathway activity, with higher scores indicating greater pathway activation. No clinical relevance threshold has been established.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom IFN scores were available at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in IFN score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 39
Change in IFN score at 16 weeks | -8.41 [-11.66 to -5.16]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.00000621, t-test, 2 sided; Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -0.84

3. Secondary Outcome: Change in Investigator's Global Assessment (IGA)
Description: The IGA is used to assess overall changes in severity across five skin conditions (alopecia areata, atopic dermatitis, vitiligo, psoriasis and hidradenitis suppurativa) scored from 0 (clear) to 4 - 5 (very severe).
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom IGA scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 42
Change in score at 16 weeks | -1.31 (0.5) [-1.76 to -0.86]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.00000061, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -0.91

4. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI)
Description: The DLQI is used to assess participant-reported impact of skin conditions on self-image, relationships, and daily activities. Possible total scores range from 0-30, with higher scores indicating a more impaired quality of life.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom DLQI scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 42
Change in score at 16 weeks | -2.88 [-3.75 to -2.01]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.00000004, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -1.03

5. Secondary Outcome: Change in Eczema Area and Severity Index (EASI) Score in Participants With Atopic Dermatitis
Description: The EASI is used to assess changes in the extent (area) and severity of atopic dermatitis (eczema). Each of four sites (head, upper limbs, trunk, and lower limbs), are weighted by overall contribution to body surface area and separately scored by using four parameters (erythema, infiltration, excoriations, lichenification), each of which is graded on a severity scale of 0 (none) to 4 (severe), as well as degree of involvement. Possible total scores range from 0-72, with higher scores indicating a more severe involvement.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom qualifying EASI scores were collected at Baseline and 16 weeks. None of the completed trial participants had qualifying EASI scores for atopic dermatitis.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Severity of Alopecia Tool (SALT) Score in Participants With Alopecia
Description: The SALT is used to assess changes in degree and extent (area) of hair loss due to alopecia areata on the head. Each of four scalp sites (left side, right side, top and back) are weighted by overall contribution to scalp surface area and rated for percent involvement. Possible total scores range from 0-72, with higher scores indicating a larger affected area.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom qualifying SALT scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 21
Change in score at 16 weeks | -28.10 [-39.27 to -16.92]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.0000393, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -1.14

7. Secondary Outcome: Change in Modified Sartorius Score (MSS) Score in Participants With Hidradenitis Suppurativa
Description: The MSS is used to assess changes in areas affected by hidradenitis suppurativa. Each of seven sites (right/left axillae, right/left groin, right/left gluteal, other) are scored by number of lesions, distance between lesions, and presence of normal skin between lesions. Possible total scores range up from 0 with no maximum, with higher scores indicating a more severe involvement.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom qualifying MSS scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 23
Change in score at 16 weeks | -19.56 [-32.19 to -6.94]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.00399, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -0.67

8. Secondary Outcome: Change in Psoriasis Area and Severity Index (PASI) Score in Participants With Psoriasis
Description: The PASI is used to assess changes in extent (area) and severity of psoriasis. Each of four sites (head, upper limbs, trunk, and lower limbs) are weighted by overall contribution to body surface area and separately scored by degree of involvement and three additional parameters (erythema, induration and desquamation), each of which is graded on a severity scale of 0 (Not severe) to 4 (very severe). Possible total scores range from 0-72, with higher scores indicating a more severe involvement.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom qualifying PASI scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 2
Change in score at 16 weeks | -7.3 [-28.90 to 14.30]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.146, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -3.04

9. Secondary Outcome: Change in Vitiligo Extent Tensity Index (VETI) in Participants With Vitiligo
Description: The VETI is used to assess changes in extent (area) of skin affected by vitiligo. Each of five sites (head, trunk, upper limbs, lower limbs, genitalia) are weighted by overall contribution to body surface area and rated for degree of de-pigmentation scale of Stage 0 (normal skin) to Stage 5 (complete de-pigmentation plus significant hair whitening) and percent involvement. Possible scores range from 0-55.5, with a higher score indicating a higher degree of involvement.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom qualifying VETI scores were collected at Baseline and 16 weeks. None of the completed trial participants had qualifying VETI scores for vitiligo.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: A Composite Cytokine Score Generated Using the Meso Scale Discovery (MSD) Platform Used to Assess Inflammatory Changes in Plasma.
Description: The Cytokine Score is a composite molecular measure used to quantify inflammatory changes. Cytokine Scores are calculated by summing standardized abundance (i.e. (abundance value - mean) / standard deviation) of a predefined panel of four inflammatory cytokines, measured in plasma samples using the Meso Scale Discovery platform. The resulting composite value provides an integrated measure of inflammatory activity, with higher scores indicating a more inflammatory state. No clinical relevance threshold has been established.
Time Frame: Baseline and 16 weeks
Population: All participants meeting medication compliance criteria and for whom Cytokine scores were collected at Baseline and 16 weeks.
Measure: Mean (95% Confidence Interval); unit: Change in score at 16 weeks
Arm/Group | On Treatment
Number analyzed (Participants) | 39
Change in score at 16 weeks | -2.15 [-2.81 to -1.49]
Statistical Analysis 1: Comparison: On Treatment; Test type: Other; p = 0.00000009, t-test, 2 sided — Two-sided paired Student t test comparing the values for each participant at Baseline and 16 weeks; Effect size (Cohen's d) = -1.05

ADVERSE EVENTS:
Time Frame: Baseline through 16 weeks.
Groups:
- On Treatment: Tofacitinib 5mg oral tablets twice daily for 16 weeks
  Tofacitinib: Treatment with oral Tofacitinib for immune-mediated skin conditions in adults with Down syndrome who completed Baseline and 16-week study time points with adequate medication compliance.
Arm/Group | On Treatment
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Treatment (N=47)
Thromboembolic event (Vascular disorders) | 1 (1) — This was a Grade 3 thromboembolic event, determined to be possibly related to the IP.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Treatment (N=47)
Grade 1 Diarrhea (Gastrointestinal disorders) | 6 (9)
Grade 2 Diarrhea (Gastrointestinal disorders) | 4 (4)
Grade 1 Vomiting (Gastrointestinal disorders) | 12 (15)
Grade 1 Rash acneiform (Skin and subcutaneous tissue disorders) | 13 (16)
Grade 1 Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (8)
Grade 2 Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (4)
Grade 2 Neutrophil count decreased (Investigations) | 3 (3)
Grade 1 Weight loss (Investigations) | 6 (7)
Grade 1 Weight gain (Investigations) | 17 (20)
Grade 2 Weight gain (Investigations) | 4 (4)
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21)
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Grade 1 Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 17 (30)
Grade 1 Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Grade 1 Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 (26)
Grade 1 Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (12)
Grade 1 Infections and infestations - COVID-19 (Infections and infestations) | 6 (6)
Grade 2 Infections and infestations - COVID-19 (Infections and infestations) | 4 (4)
Grade 1 Skin infection (Infections and infestations) | 4 (4)
Grade 1 Fever (General disorders) | 7 (11)
Grade 1 Fatigue (General disorders) | 7 (10)
Grade 1 Headache (Nervous system disorders) | 4 (6)
Grade 1 Stomach pain (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT04246372/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04246372/ICF_002.pdf